CLINICAL TRIAL: NCT01341392
Title: A Randomized, Open-label, Multiple Dose, Three-treatment, Three-period, Six-sequence Crossover Clinical Trial to Investigate the Pharmacokinetic Drug Interaction Between CKD-501 and Amlodipine After Oral Administration in Healthy Male Volunteers
Brief Title: Drug-drug Interaction Study(CKD-501, Amlodipine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Severance Hospital (Other)
Responsible Party: Chin Kim, Chong Kun Dang Pharmaceutical
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19HPS11H
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Drug-Drug interaction between the CKD-501 and Amlodipine
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CKD-501 0.5mg (Experimental): Subjects received CKD-501 0.5mg once daily for 10 days. Subjects received amlodipine 10mg once daily for 10 days. Subjects received CKD-501 0.5mg and amlodipine 10mg for 10 days.
  Interventions: Drug: CKD-501
- CKD-501 Amlodipine (Experimental): Subjects received CKD-501 0.5mg once daily for 10 days. Subjects received amlodipine 10mg once daily for 10 days. Subjects received CKD-501 0.5mg and amlodipine 10mg for 10 days.
  Interventions: Drug: CKD-501 amlodipine
- Amlodipine 10mg (Experimental): Subjects received CKD-501 0.5mg once daily for 10 days. Subjects received amlodipine 10mg once daily for 10 days. Subjects received CKD-501 0.5mg and amlodipine 10mg for 10 days.
  Interventions: Drug: amlodiopine

INTERVENTIONS:
Drug: CKD-501 — Subjects received CKD-501 0.5mg once daily for 10 days. Subjects received amlodipine 10mg once daily for 10 days. Subjects received CKD-501 0.5mg and amlodipine 10mg for 10 days.
  Other Names: Lobeglitazone
  Arms: CKD-501 0.5mg
Drug: amlodiopine — Subjects received CKD-501 0.5mg once daily for 10 days. Subjects received amlodipine 10mg once daily for 10 days. Subjects received CKD-501 0.5mg and amlodipine 10mg for 10 days.
  Arms: Amlodipine 10mg
Drug: CKD-501 amlodipine — Subjects received CKD-501 0.5mg once daily for 10 days. Subjects received amlodipine 10mg once daily for 10 days. Subjects received CKD-501 0.5mg and amlodipine 10mg for 10 days.
  Arms: CKD-501 Amlodipine

SUMMARY:
The purpose of this study is to assess the pharmacokinetic drug interaction between CKD-501 and amlodipine after oral administration in healthy male volunteers.

DETAILED DESCRIPTION:
Volunteers doses three times over the period of CKD-501 0.5mg or Amlodipine 10mg alone/co-administrate, repeated doses are 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 45 years old in healthy males
* Body weight ≥ 55kg and 18.5 ≤ IBW < 25
* Agreement with written informed consent

Exclusion Criteria:

* Subject has a history affects the ADME of drug
* Hypersensitivity reactions to drugs or clinically significant hypersensitivity reactions in the history of party
* Inadequate subject by medical examination(medical history, physical examination, ECG, laboratory test)
* AST,ALT > UNL * 1.25 or Total bilirubin > UNL * 1.5
* Estimated GFR(MDRD) < 80
* SBP >150 mmHg, SBP < 100 mmHg or DBP > 100 mmHg, DBP < 60 mmHg or Pulse > 100 per/min, Pulse < 50 per/min
* Substance abuse, or a history of drug abuse showed a positive for the party
* Continued to be taking caffeine (caffeine > 5 cup/day), drinking (alcohol > 210 g/week) or cannot stop drinking or severe heavy smoker(cigarette > 10 cigarettes per day)during clinical trials
* Medication with drug-mediated induction/inhibition metabolic enzyme within 30 days or with may affect the clinical trial
* Medication within 2 weeks in the first professional medical, medicine, OTC, vitamins taking
* Subject takes grapefruit within 1 month
* Previously participated in other trial within 60 days
* Previously donate whole blood within 60 days or component blood within 30 days
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
CKD-501 AUC | Pre dose(D8-9, D29-30, D50-51), 0, 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24hr
Amlodipine AUC | Pre dose(D8-9, D29-30, D50-51), 0, 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 48, 72hr

SECONDARY OUTCOMES:
CKD-5011 Tmax | Pre dose(D8-9, D29-30, D50-51), 0, 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24hr
Amlodipine Tmax | Pre dose(D8-9, D29-30, D50-51), 0, 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 7, 8, 10, 12, 16, 24, 48, 72hr

CONTACTS AND LOCATIONS:
Overall Officials: Minsoo Park, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim CO, Sil Oh E, Kim C, Park MS. Pharmacokinetic Interaction Between Amlodipine and Lobeglitazone, a Novel Peroxisome Proliferator-activated Receptor-gamma Agonist, in Healthy Subjects. Clin Ther. 2015 Sep;37(9):1999-2006.e1. doi: 10.1016/j.clinthera.2015.06.009. Epub 2015 Jul 7. PMID 26163202